CLINICAL TRIAL: NCT05519670
Title: A Phase 1b/2 Trial Evaluating Safety and Efficacy of CAPecitabine in Combination With Ni-rapaRIb in HER2-negative Advanced Breast canCEr
Acronym: CAPRICE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPRICE-IPC 2020-053
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Only Arm (Experimental): niraparib + capecitabine treatment
  Interventions: Drug: Niraparib Oral Product

INTERVENTIONS:
Drug: Niraparib Oral Product — Niraparib + capecitabine treatment

SUMMARY:
This study will be to combine oral capecitabine and oral niraparib such thz association may increase clinical benefits of PARP inhibitors in germline BRCA mutated HER2 negative advanced breast cancer patients.

DETAILED DESCRIPTION:
In spite of multimodal treatment, prognosis of HER2 negative metastatic breast cancers remains poor and innovative targeted therapeutic approaches are urgently warranted. While PARP inhibi-tors as single agent have demonstrated moderate improvement in progression-free survival and quality of life in pre-treated HER2 negative advanced breast cancer patients with germline BRCA mutation, they failed to improve overall survival in this setting. In addition, most of clinical trials testing combinations of chemotherapy and PARP inhibitors have been limited by overlapping hematological toxicities, or have used low dosage PARP inhibitors with short exposure time and with uncertain benefits. The therapeutic strategy selected in this study will be to combine oral capecitabine (2 weeks on, 1 week off, as recommended in monotherapy) and oral niraparib (con-tinuously for a cycle of 21 days). Such an association may increase clinical benefits of PARP inhibitors in germline BRCA mutated HER2 negative advanced breast cancer patients, while po-tentially expanding clinical interest of PARP inhibitors in patients without germline BRCA muta-tion (either with or without HRD).

ELIGIBILITY:
Inclusion Criteria:

1. Women or men aged 18 or more
2. Histologically-confirmed advanced breast cancer (metastatic or locally advanced)
3. Tumor without overexpression of HER2 (HER2 1+ in IHC, or IHC 2+ and FISH/ CISH negative) in samples from the primary and/or secondary tumor
4. Hormone receptor status known
5. Endocrine insensitive (hormone receptor negative or Endocrine (aromatase inhibitor)-resistant (a CDK4/6-based endocrine treatment must have been administered as a first-line of second-line treatment, unless primary endocrine-refractory disease as defined as relapse within the first 2 years of aromatase-based adjuvant endocrine therapy or progression under endocrine treatment administered for metastatic disease within 6 months of initiation))
6. Progressive disease patients who are eligible to a treatment with capecitabine: after fail-ure to taxanes and anthracycline-based chemotherapy (unless contraindicated) (neoadjuvant, adjuvant or metastatic setting)
7. A representative tumor specimen must be available for molecular testing. An archival tu-mor sample may be submitted (<6 months); however, if one is not available, a newly obtained tumor biopsy specimen must be submitted instead
8. Measurable disease according to RECIST1.1
9. Symptomatic, untreated, or actively progressing central nervous system (CNS) metasta-ses are not eligible. Patients with a history of treated CNS lesions are eligible, provided all of the following criteria are met:

   1. Measurable or non-measurable disease, per RECIST v. 1.1, must be present outside the CNS
   2. No history of intracranial haemorrhage or spinal cord haemorrhage
   3. Metastases are limited to the cerebellum or the supratentorial region (i.e., no metasta-ses to the midbrain, pons, medulla, or spinal cord).
   4. There is no evidence of interim progression between completion of CNS-directed ther-apy and the screening brain scan.
   5. The patient has not received stereotactic radiotherapy within 7 days prior to initiation of study treatment or whole-brain radiotherapy within 14 days prior to initiation of study treatment.
   6. The patient has no ongoing requirement for corticosteroids as therapy for CNS disease. Anticonvulsant therapy at a stable dose is permitted.

Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan.

10. Patients must have an estimated survival of at least 3 months 11. WHO performance status (ECOG) from 0 to 1 12. Adequate hematological and coagulation function: Hb ≥ 10.0 g/dL, ANC ≥ 1500/mm3 platelets ≥ 150 000/mm3, INR ≤ 1.5 13. Adequate hepatic function : total serum bilirubin ≤ 1x ULN, or total bilirubin ≤ 2.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert's Syndrome, ALAT and ASAT ≤ 1.5 x ULN 14. Adequate renal function: serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60mL/min 15. Adequate ionic balance: potassium, calcium (corrected for serum albumin), magnesium, sodium and phosphorus within normal limits for the institution 16. Participant must have normal blood pressure or adequately treated and controlled hyperten-sion17. A female participant is eligible if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

* Is not a woman of childbearing potential (WOCBP) OR
* Is a WOCBP and must agree to use a highly effective contraceptive method (described in 6.6.2) while on treatment and for at least 180 days after study drugs discontinuation.

  18. A WOCBP must have a negative pregnancy test (highly sensitive urine test or serum test as required by local regulations) within 72 hours before the first dose of study treatment.

  19. Male participants are eligible to participate if they agree to the following during the interven-tion period and for at least 90 days after the last dose of study treatment:
* Refrain from donating sperm
* Must agree to use a male condom (and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak) 20. Patient must be affiliated to a Social Security system 21. Patient information and written informed consent form signed 22. Must be able to swallow and retain orally administered study treatment. 23. For expansion cohort: inclusion will be done regarding availability of homologous recom-bination status

Exclusion Criteria:

1. Prior treatment with a PARP inhibitor and capecitabine for metastatic disease, (Patients treat-ed with these drugs in the adjuvant setting are allowed to participate if they experienced 2 years from end of treatment and metastatic relapse)
2. Patient has a Dihydropyrimidine dehydrogenase deficiency (DPD)
3. Patients must not have received anticancer chemotherapy, targeted therapy within 2 weeks prior of the study. Endocrine therapy must have been discontinued 7 or more days before Cycle 1 Day 1. Participant must not have had investigational therapy administered within 4 weeks or with-in a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study.
4. Palliative radiotherapy must have been completed 14 or more days before Cycle 1 Day 1. Biphosphonates and denosumab are allowed.
5. Major surgery within 3 weeks prior to registration. Patients must have recovered from earlier major surgery before registration.
6. Persistent toxicities (≥NCI-CTCAE grade 2) caused by previous cancer therapy, excluding alopecia and NCI-CTCAE grade 2 peripheral neuropathy.
7. Immunocompromised patients (e.g. HIV) for part I and but patients with well controlled HIV could be included in part II (negative viral load)
8. Patients considered at poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection, symptomatic congestive heart fail-ure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, or Posterior Reversible Encephalopathy Syn-drome (PRES).
9. Mean resting QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 consecutive electrocardiograms using Fridericia's Correction.
10. Active or prior documented inflammatory bowel disease (Crohn's disease, ulcerative colitis).
11. Patients unable to swallow orally administered medication, patients with gastrointestinal dis-orders likely to interfere with absorption of niraparib, and patients with long-term oral anticoagu-lant therapy.
12. Pregnant or breast-feeding women. Participant must agree to not breastfeed during the study and for 30 days after the last dose of study treatment
13. Known hypersensitivity to niraparib or capecitabine or any of the excipients of the products
14. Patient is currently receiving or has received sorivudine or brivudine within 4 weeks prior to starting capecitabine
15. Patient has received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy
16. Patient has received colony-stimulating factors (e.g. granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) ≤ 4 weeks prior to initiating protocol therapy
17. Patient has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks
18. Patient has any known history of myelodysplastic syndrome (MDS) or acute myeloid leuke-mia (AML)
19. Patient has a diagnosis, detection, or treatment of another type of cancer ≤ 2 years prior to initiating study therapy with the following exceptions: basal or squamous cell carcinoma of the skin, cervical cancer in situ that has been definitively treated, adequately treated nonmelanoma skin cancer, ductal carcinoma in situ (DCIS) of the breast.
20. Patient has known active hepatitis B (e.g. hepatitis B surface antigen (HBsAg] reaction) or hepatitis C (e.g. hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected)
21. Participants have received live vaccine within 30 days of planned start of study registration. 22. Participants have current active pneumonitis or any history of pneumonitis requiring steroids (any dose) or immunomodulatory treatment within 90 days of planned start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities (DLT) | 3 weeks
  incidence of Dose-Limiting Toxicities (DLT)
efficacy with objective response rate (ORR) | 6 months
  rate of patients experiencing an objective response

SECONDARY OUTCOMES:
adverse events | 6 months
  incidence of adverse events
Pharmacokinetics (PK) | 15 days
  Plasma concentrations and basic PK parameters of niraparib and capecitabine when adminis-tered in combination

IPD SHARING:
Plan to Share IPD: No